CLINICAL TRIAL: NCT04349098
Title: A Phase 2 Randomized Single-Blind Study to Evaluate the Activity and Safety of Low Dose Oral Selinexor (KPT-330) in Patients With Severe COVID-19 Infection
Brief Title: Evaluation of Activity and Safety of Oral Selinexor in Participants With Severe COVID-19 Infection
Acronym: Coronavirus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XPORT-CoV-1001; 2020-001411-25 (EudraCT Number)
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — selinexor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Selinexor 20 mg (Experimental): Participants will receive 20 milligram (mg) of selinexor oral tablet on Days 1, 3, and 5 of each week for up to 2 weeks (14 days). If the participant is tolerating therapy and clinically benefitting, dosing can continue for an additional 2 weeks (28 days).
  Interventions: Drug: Selinexor
- Placebo (Placebo Comparator): Participants will receive 20 mg of placebo matched to selinexor oral tablet on Days 1, 3, and 5 of each week for up to 2 weeks (14 days). If the participant is tolerating therapy and clinically benefitting, dosing can continue for an additional 2 weeks (28 days).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Selinexor — Participants will receive 20 mg of selinexor.
  Other Names: KPT-330; XPOVIO
  Arms: Selinexor 20 mg
Other: Placebo — Participants will receive 20 mg of placebo matched to selinexor.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the activity of low dose oral selinexor (KPT-330) and to evaluate the clinical recovery, the viral load, length of hospitalization and the rate of morbidity and mortality in participants with severe COVID-19 compared to placebo. The study had 2 arms and evaluated selinexor 20 mg + standard of care (SoC) and placebo + SoC. As the treatment for COVID-19 is rapidly evolving, the SoC varied over time and across regions of the world.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed laboratory diagnosis of SARS-CoV2 by standard FDA-approved reverse transcription polymerase chain reaction (RT-PCR) assay or equivalent FDA-approved testing (local labs).
* Currently hospitalized.
* Informed consent provided as above (it is recommended that participants are dosed with study drug within 12 hours of consent).
* Has symptoms of severe COVID-19 as demonstrated by:

  * At least one of the following: fever, cough, sore throat, malaise, headache, muscle pain, shortness of breath at rest or with exertion, confusion, or symptoms of severe lower respiratory symptoms including dyspnea at rest or respiratory distress.
  * Clinical signs indicative of lower respiratory infection with COVID-19, with at least one of the following: SaO2 <92% on room air in last 12 hours or requires > 4 liters per minute (LPM) oxygen by nasal canula, non-rebreather/Ventimask or high flow nasal canula in order maintain SaO2 ≥92%, PaO2/FiO2 <300 millimeter per mercury (mm/hg).
* Elevated C-reactive protein (CRP) > 2 x upper limit of normal (ULN).
* Concurrent anti-viral and/or anti-inflammatory agents (e.g., biologics, hydroxychloroquine) are permitted. If in the physician's judgment, it is in the best interest of the participant to use anti-viral or anti-inflammatory treatments, these treatments are to be documented in the participant's chart and entered in the electronic case report form.
* Female participants of childbearing potential must have a negative serum pregnancy test at Screening. Female participants of childbearing potential and fertile male participants must use highly effective methods of contraception throughout the study and for 3 months following the last dose of study treatment.

Exclusion Criteria:

* Evidence of critical COVID-19 based on:

  * Respiratory failure (defined by endotracheal intubation and mechanical ventilation, oxygen delivered by noninvasive positive pressure ventilation, or clinical diagnosis of respiratory failure in setting of resource limitations)
  * Septic shock (defined by Systolic blood pressure [BP] < 90 mm Hg, or Diastolic BP < 60 mm Hg)
  * Multiple organ dysfunction/failure
* In the opinion of the investigator, unlikely to survive for at least 48 hours from screening or anticipate mechanical ventilation within 48 hours.
* Inadequate hematologic parameters as indicated by the following labs:

  * Participants with severe neutropenia (ANC <1000 x 10^9/L) or
  * Thrombocytopenia (e.g., platelets <100,000 per microliter of blood)
* Inadequate renal and liver function as indicated by the following labs:

  * Creatinine clearance (CrCL) <20 mL/min using the formula of Cockcroft and Gault
  * Aspartate transaminase (AST) or alanine transaminase (ALT) > 5 x ULN
* Hyponatremia defined as sodium < 135 milliequivalents per liter (mEq/L).
* Unable to take oral medication when informed consent is obtained.
* Participants with a legal guardian or who are incarcerated.
* Treatment with strong CYP3A inhibitors or inducers.
* Pregnant and breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (20):
  - UCLA, Los Angeles, California
  - Kaiser Permanente Oakland, Oakland, California
  - UC Davis Health, Sacramento, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Kaiser Permanente San Francisco, San Francisco, California
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Healthcare, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - Karmanos, Detroit, Michigan
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Michigan Center of Medical Research, Royal Oak, Michigan
  - Columbia University, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute-Atrium Health University City, Charlotte, North Carolina
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Baylor Scott & White Dallas, Dallas, Texas
  - MultiCare Institute for Research & Innovation (Puget Sound), Tacoma, Washington
- Hospital Hietzing, 2. Medical department - Center for Diagnosis and Therapy of Rheumatic Diseases, Vienna, Austria
- France (3):
  - CHU Bordeaux, Bordeaux
  - CHU Lyon, Lyon
  - CHU Nantes, Nantes
- Israel (3):
  - Hadassah MC, Jerusalem
  - Hasharon Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Servicio de Medicina Interna, Hospital Universitario de Salamanca, Universidad de Salamanca, Salamanca
- United Kingdom (4):
  - Princess Royal University Hospital, Kent
  - Kings College Hospital, London
  - The Royal Marsden Hospital, London
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 20 sites in the United States of America,1 site in Austria, 3 sites in France and Israel, 2 sites in Spain, and 4 sites in the United Kingdom from 17 Apr 2020 to 05 Oct 2020.
Pre-assignment Details: A total of 190 participants were enrolled and randomized, of which 188 participants received study treatment in this study.
Groups:
- Selinexor 20 mg: Participants received a single dose of Selinexor 20 milligrams (mg) tablets orally on Days 1, 3 and 5 of each week for up to 2 weeks. The participant tolerated therapy and showed clinical benefit, dosing continued for an additional 2 weeks (on Days 15, 17, 19, 22, 24, and 26).
- Placebo: Participants received a single dose of placebo matched to selinexor tablets orally on Days 1, 3 and 5 of each week for up to 2 weeks. The participant tolerated therapy and showed clinical benefit, dosing continued for an additional 2 weeks (on Days 15, 17, 19, 22, 24, and 26).
Period: Overall Study
Arm/Group | Selinexor 20 mg | Placebo
Started | 103 | 87
Treated | 102 | 86
Completed | 65 | 61
Not Completed | 38 | 26
Not completed — Death | 16 | 8
Not completed — Lost to Follow-up | 11 | 8
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Other | 3 | 5

BASELINE CHARACTERISTICS:
Population: PV 1-6 population included participants randomized into the study under protocol versions 1-6.
Groups:
- Total: Total of all reporting groups
Arm/Group | Selinexor 20 mg | Placebo | Total
Number analyzed (Participants) | 103 | 87 | 190
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (16.12) | 56.5 (14.64) | 56.5 (15.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 60 | 48 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 32 | 73
  Not Hispanic or Latino | 59 | 53 | 112
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 23 | 24 | 47
  White | 44 | 34 | 78
  More than one race | 19 | 14 | 33
  Unknown or Not Reported | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At-least a 2-Point Improvement in Ordinal Scale
Description: Ordinal Scale 2-Point improvement was defined as percentage of participants with at least a 2-points improvement (increase from baseline) by Day 14. Baseline score was defined as the last score measured before first dosing. The 8-point ordinal scale ranges from 1 to 8: where 1= death, 2= hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3= hospitalized, on non-invasive ventilation or high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (coronavirus disease 2019 [COVID-19] related or otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7= not hospitalized, limitation on activities and/or requiring home oxygen; 8= not hospitalized, no limitations on activities.
Time Frame: Baseline up to Day 14
Population: The intent-to-treat (ITT) population included all participants who were randomized in the study with confirmed severe acute respiratory syndrome coronavirus (SARS-CoV2) infection under protocol version (PV) 6.0 and above, regardless of whether or not they receive study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 66 | 51
Percentage of participants | 60.6 [47.8 to 72.4] | 60.8 [46.1 to 74.2]
Statistical Analysis 1: Comparison: Selinexor 20 mg vs Placebo; Test type: Superiority; p = 0.6750, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.39 to 1.79]

2. Secondary Outcome: Percentage of Participants With at Least a 2-Point Improvement in the Ordinal Scale up to Day 7
Description: Ordinal Scale 2-points improvement was defined as percentage of participants with at least a 2-points improvement (increase from baseline) by Day 7. Baseline score was defined as the last score measured before first dosing. The 8-point ordinal scale ranges from 1 to 8: where, 1= death, 2= hospitalized, on invasive mechanical ventilation or ECMO; 3= hospitalized, on non-invasive ventilation or high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7= not hospitalized, limitation on activities and/or requiring home oxygen; 8= not hospitalized, no limitations on activities.
Time Frame: Baseline up to Day 7
Population: PV 1-6 population included participants randomized into the study under protocol versions 1-6.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 103 | 87
Percentage of participants | 30.1 [21.5 to 39.9] | 32.2 [22.6 to 43.1]

3. Secondary Outcome: Percentage of Participants With at Least a 1-Point Improvement in the Ordinal Scale
Description: Ordinal Scale 1-point improvement was defined as percentage of participants with at least 1-point improvement (increase from baseline) by Day 7 and 14. Baseline score was defined as the last score measured before first dosing. The 8-point ordinal scale ranges from 1 to 8: where 1= death, 2= hospitalized, on invasive mechanical ventilation or ECMO; 3= hospitalized, on non-invasive ventilation or high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7= not hospitalized, limitation on activities and/or requiring home oxygen; 8= not hospitalized, no limitations on activities.
Time Frame: Baseline up to Day 7 and 14
Population: PV 1-6 population included participants randomized into the study under protocol versions 1-6.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 103 | 87
Percentage of participants
  Day 7 | 51.5 [41.4 to 61.4] | 50.6 [39.6 to 61.5]
  Day 14 | 72.8 [63.2 to 81.1] | 72.4 [61.8 to 81.5]

4. Secondary Outcome: Time to Clinical Improvement of 2-points Using Ordinal Scale (TTCI-2)
Description: TTCI-2 was defined as the time from randomization to an improvement of 2-points using 8-points Ordinal Scale. The 8-point ordinal scale ranges from 1 to 8: where 1= death, 2= hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3= hospitalized, on non-invasive ventilation or high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (coronavirus disease 2019 [COVID-19] related or otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7= not hospitalized, limitation on activities and/or requiring home oxygen; 8= not hospitalized, no limitations on activities.
Time Frame: Baseline up to Day 28
Population: ITT Population included all participants who were randomized in the study with confirmed SARS-CoV2 infection under protocol version 6.0 and above, regardless of whether or not they receive study treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 66 | 51
Days | 10.0 [8.0 to 14.0] | 10.0 [8.0 to 14.0]

5. Secondary Outcome: Overall Death Rate
Description: Overall death rate was defined as the percentage of participants who died on or before Day 28.
Time Frame: Baseline up to Day 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 66 | 51
Percentage of participants | 15.2 [7.5 to 26.1] | 3.9 [0.5 to 13.5]

6. Secondary Outcome: Rate of Mechanical Ventilation (RMV)
Description: The rate of RMV was defined as the percentage of participants who ever used invasive mechanical ventilation or ECMO during the hospital stay.
Time Frame: Baseline up to Day 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 66 | 51
Percentage of participants | 13.6 [6.4 to 24.3] | 11.8 [4.4 to 23.9]

7. Secondary Outcome: Rate of Intensive Care Unit (ICU) Admission
Description: The rate of ICU admission was defined as the percentage of participants with ICU admissions.
Time Frame: Baseline up to Day 28
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 66 | 51
Percentage of participants | 48.5 [36.0 to 61.1] | 41.2 [27.6 to 55.8]

8. Secondary Outcome: Length of Hospitalization
Description: Length of hospitalization (days) was defined as (first hospital discharge date - date of randomization + 1).
Time Frame: Baseline up to Day 67
Population: as for outcome 4
Measure: Median (Full Range); unit: Days
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 66 | 51
Days | 9.0 [3 to 39] | 9.0 [3 to 67]

9. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Levels
Description: The anti-inflammatory and immune effects of selinexor were assessed by CRP levels. Baseline was defined as the most recent non-missing measurement prior to the first administration of study treatment. Change from Baseline at the indicated time points was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline, Day 3, 5, 8, 12, 15, 19, 22 and 26
Population: PV 1-6 population included participants randomized into the study under protocol versions 1-6. Here, "Number Analyzed" signified those participants who were evaluable for this outcome measure at a specified time-point.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 103 | 87
milligram per liter (mg/L)
  Change at Day 3: number analyzed (Participants) | 88 | 74
  Change at Day 3 | -47.9660 (99.06082) | -42.9658 (89.09341)
  Change at Day 5: number analyzed (Participants) | 83 | 69
  Change at Day 5 | -74.4735 (114.52388) | -68.6191 (108.19671)
  Change at Day 8: number analyzed (Participants) | 57 | 45
  Change at Day 8 | -83.3460 (93.83500) | -74.4669 (117.66505)
  Change at Day 12: number analyzed (Participants) | 31 | 27
  Change at Day 12 | -86.9158 (123.54705) | -93.2744 (131.56709)
  Change at Day 15: number analyzed (Participants) | 10 | 15
  Change at Day 15 | -87.9800 (121.19999) | -98.7940 (87.65276)
  Change at Day 19: number analyzed (Participants) | 7 | 9
  Change at Day 19 | -66.2143 (86.55049) | -124.3233 (102.04161)
  Change at Day 22: number analyzed (Participants) | 10 | 5
  Change at Day 22 | -90.7100 (149.25579) | -47.5620 (171.49171)
  Change at Day 26: number analyzed (Participants) | 5 | 5
  Change at Day 26 | -37.2800 (141.41390) | -129.5020 (46.26178)

10. Secondary Outcome: Change From Baseline in Ferritin Levels
Description: The anti-inflammatory and immune effects of selinexor were assessed by ferritin levels. Baseline was defined as the most recent non-missing measurement prior to the first administration of study treatment. Change from Baseline at the indicated time points was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline, Day 3, 5, 8, 12, 15, 19, 22 and 26
Population: PV 1-6 population included participants randomized into the study under protocol versions 1-6. Here, "Number Analyzed" signified those participants who were evaluable for this outcome measure at a specified timepoint.
Measure: Mean (Standard Deviation); unit: microgram/liter (mcg/L)
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 103 | 87
microgram/liter (mcg/L)
  Change at Day 3: number analyzed (Participants) | 82 | 70
  Change at Day 3 | 80.8415 (759.10075) | -61.9843 (542.09460)
  Change at Day 5: number analyzed (Participants) | 79 | 63
  Change at Day 5 | -25.7000 (856.16619) | -155.3111 (773.76777)
  Change at Day 8: number analyzed (Participants) | 53 | 39
  Change at Day 8 | 226.6113 (1673.46162) | -292.2462 (738.07874)
  Change at Day 12: number analyzed (Participants) | 29 | 25
  Change at Day 12 | 193.5793 (1203.33385) | -352.5280 (741.13673)
  Change at Day 15: number analyzed (Participants) | 10 | 14
  Change at Day 15 | 204.3900 (557.29217) | -356.8429 (476.04151)
  Change at Day 19: number analyzed (Participants) | 6 | 8
  Change at Day 19 | -15.9333 (462.40358) | -231.2374 (599.98919)
  Change at Day 22: number analyzed (Participants) | 10 | 4
  Change at Day 22 | -103.9900 (636.89555) | -102.0000 (417.51247)
  Change at Day 26: number analyzed (Participants) | 6 | 4
  Change at Day 26 | -150.1167 (535.94141) | -25.7500 (231.43232)

11. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH) Levels
Description: The anti-inflammatory and immune effects of selinexor were assessed by LDH levels. Baseline was defined as the most recent non-missing measurement prior to the first administration of study treatment. Change from Baseline at the indicated time points was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline, Day 3, 5, 8, 12, 15, 19, 22 and 26
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units/liter (U/L)
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 103 | 87
units/liter (U/L)
  Change at Day 3: number analyzed (Participants) | 76 | 63
  Change at Day 3 | -13.86 (148.231) | -11.86 (151.630)
  Change at Day 5: number analyzed (Participants) | 74 | 62
  Change at Day 5 | -49.12 (175.722) | 31.85 (326.281)
  Change at Day 8: number analyzed (Participants) | 52 | 40
  Change at Day 8 | -75.85 (264.840) | -10.93 (166.876)
  Change at Day 12: number analyzed (Participants) | 28 | 25
  Change at Day 12 | -107.39 (198.092) | -16.84 (232.605)
  Change at Day 15: number analyzed (Participants) | 11 | 14
  Change at Day 15 | -71.82 (193.543) | -51.50 (148.063)
  Change at Day 19: number analyzed (Participants) | 8 | 7
  Change at Day 19 | -96.38 (200.164) | -74.14 (114.271)
  Change at Day 22: number analyzed (Participants) | 10 | 5
  Change at Day 22 | -129.70 (177.454) | -75.40 (43.569)
  Change at Day 26: number analyzed (Participants) | 6 | 4
  Change at Day 26 | -169.50 (213.481) | 4.50 (130.733)

12. Secondary Outcome: Changes From Baseline in Blood Plasma Cytokines Levels-Interleukin-6 (IL-6)
Description: The anti-inflammatory and immune effects of selinexor were assessed by blood plasma cytokines like IL-6. Baseline was defined as the most recent non-missing measurement prior to the first administration of study treatment. Change from Baseline at the indicated time points was calculated as the value at the indicated time points minus the value at Baseline.
Time Frame: Baseline, Day 3, 5, 8, 12, 15, 22 and 26
Population: PV 1-6 population included participants randomized into the study under protocol versions 1-6. Here, Overall Number of participants analyzed included all participants with baseline data and "Number Analyzed" signified those participants who were evaluable for this outcome measure at a specified time-point.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 103 | 87
nanograms/milliliter (ng/mL)
  Change at Day 3: number analyzed (Participants) | 38 | 23
  Change at Day 3 | -19.931 (51.2072) | 2.046 (49.0258)
  Change at Day 5: number analyzed (Participants) | 38 | 26
  Change at Day 5 | -10.786 (102.9160) | -77.509 (408.0085)
  Change at Day 8: number analyzed (Participants) | 28 | 15
  Change at Day 8 | -13.909 (161.6803) | 183.728 (662.7908)
  Change at Day 12: number analyzed (Participants) | 13 | 9
  Change at Day 12 | 276.289 (1541.3692) | 223.637 (715.5904)
  Change at Day 15: number analyzed (Participants) | 4 | 4
  Change at Day 15 | -34.850 (28.6357) | 207.625 (408.5783)
  Change at Day 22: number analyzed (Participants) | 3 | 0
  Change at Day 22 | -8.600 (11.8072) |
  Change at Day 26: number analyzed (Participants) | 1 | 0
  Change at Day 26 | -23.400 |

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Adverse events are defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs are defined as those AEs that develop or worsen after the first dose of study drug. TEAEs included both Serious and non-serious TEAEs.
Time Frame: From start of study drug administration up to Day 58
Population: All-treat population consisted of the subset of ITT participants who took at least one dose of study treatment on this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor 20 mg | Placebo
Number analyzed (Participants) | 102 | 86
Participants
  Participants with TEAEs | 75 | 49
  Participants with Serious TEAEs | 23 | 14

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Day 58
Description: All-treat population consisted of the subset of ITT participants who took at least one dose of study treatment on this study.
Arm/Group | Selinexor 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 16/102 | 8/86
Serious Adverse Events (participants affected / at risk) | 23/102 | 14/86
Other Adverse Events (participants affected / at risk) | 69/102 | 45/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor 20 mg (N=102) | Placebo (N=86)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Long QT syndrome (Cardiac disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 2
Systemic inflammatory response syndrome (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Viral myocarditis (Infections and infestations) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Catatonia (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor 20 mg (N=102) | Placebo (N=86)
Anaemia (Blood and lymphatic system disorders) | 9 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 2
Leukopenia (Blood and lymphatic system disorders) | 5 | 1
Constipation (Gastrointestinal disorders) | 14 | 9
Nausea (Gastrointestinal disorders) | 13 | 6
Diarrhoea (Gastrointestinal disorders) | 10 | 4
COVID-19 (Infections and infestations) | 5 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 7
Alanine aminotransferase increased (Investigations) | 8 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 24 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Hypotension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT04349098/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/98/NCT04349098/SAP_001.pdf